CLINICAL TRIAL: NCT02982265
Title: "Pre-eclampsia/Eclampsia in Italy Over the Years 2010-2016" Retrospective Observational Multicenter Study Carried Out Through an On-line Self-administered Questionnaire
Brief Title: Pre-eclampsia/Eclampsia in Italy Over the Years 2010-2016
Status: Completed | Type: Observational
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Chiara Viviani, Dr, Papa Giovanni XXIII Hospital
Other Study IDs: Reg. 2016/0161
Record Dates: First submitted 2016-11-14; First posted 2016-12-05 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Preeclampsia/Eclampsia
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Pre-eclampsia is a heterogeneous multisystem disorder that complicates 2-8% of pregnancies and remains a leading cause of maternal and perinatal mortality and morbidity.

Pre-eclampsia is defined as new onset of hypertension (defined as a diastolic blood pressure ≥ 90 mm Hg and a systolic blood pressure ≥ 140 mmHg on at least two different recordings taken at least 4-6 h apart and less than 7 days apart, using an appropriate cuff) and substantial proteinuria (defined as excretion of protein ≥300 mg in 24 h or a protein concentration ≥ 300 mg/L or ≥ "1 +" on dipstick in at least two random urine samples taken at least 4-6 h apart but no more than 7 days apart) at or after 20 weeks of gestation.

Pre-eclampsia only occurs in the presence of placenta and is resolved by delivery of the same. However, the underlying causes of the disease remain largely unknown.

DETAILED DESCRIPTION:
Poor placentation is considered a powerful predisposing factor for pre-eclampsia. Recently, it has been suggested that the occurrence of pre-eclampsia requires a combination of an excessive or atypical maternal immune response to the trophoblast and/or exaggerated endothelial activation as well as a generalised hyper-inflammatory state resulting in endothelial dysfunction and associated increased vascular reactivity. Any factors (maternal and paternal constitutional, genetic and environmental risk factors) that enhance these responses would predispose to pre-eclampsia.

The list of predisposing factors includes: extremes of maternal age, black race, previous history of pre-eclampsia, family history of pre-eclampsia, multifetal gestation, ≥ 10 years from previous pregnancy, limited sperm exposure, first paternity, pregnancies after donor insemination (assisted reproductive technology), oocyte donation or embryo donation, chronic hypertension or renal disease, rheumatic disease, maternal low birth weight, obesity and insulin resistance, pre-gestational diabetes mellitus, increased testosterone, increased homocysteine concentration, atherosclerosis (increased triglycerides and LDL, decreased HDL), maternal infections, pre-existing thrombophilia, maternal susceptibility genes and hydropic degeneration of placenta. Finally, smoking seems to be inversely correlated with pre-eclampsia.

Pre-eclampsia can result in a fetal syndrome characterized by fetal growth restriction, reduced amniotic fluid, abnormal oxygenation, fetal demise and preterm birth. Moreover, women with pre-eclampsia are at increased risk for abruptio placentae, disseminated coagulopathy/HELLP syndrome, pulmonary oedema, acute renal failure, eclampsia, cerebral haemorrhage, death and cardiovascular or renal disease.

Early prediction of pre-eclampsia would allow for close surveillance and preventive strategies

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand the Italian language and fill in the questionnaire, including access to the Internet.
* Ability of both parents to give informed consent to the processing of personal data, with the understanding that the consent could be withdrawn at any time

Exclusion Criteria:

* Inability to reach the patients by telephone and inform them about the study
* Death or incapacitating illness of one or both parents following discharge from hospital
* Refusal of one or both parents to disclose their email address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Women discharged from the enrolling Centres with a diagnosis of preeclampsia and/or eclampsia over the years 2010-2016, identified by the ICD-9-CM codes 642.4 to 642.44, 642.5 to 642.54, 642.6 to 642.64 and 642.7 to 642.74.
  * Fathers
Sampling Method: Non-Probability Sample
Enrollment: 1527 (Actual)
Dates: Start 2016-08; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Incidence of preeclampsia/eclampsia in Italy | Three months
Aggregation of predisposing factors to pre-eclampsia / eclampsia in Italy measured by a novel multiple choice on-line questionnaire | Three months
  Either, or maternal and paternal: extremes of age (years), extremes of weight (BMI in kg/m2), blood group, ethnic group, level of education (primary, secondary or academic), cardiovascular predisposing factors (hypertension defined as over 140/90 mmHg BP, diabetes mellitus defined as fasting glycemia over 126 mg/dl or over 200mg/dl in a glucose tolerance test, hypercholesterolemia defined as LDL over 240mg/dl, hyperhomocysteinemia defined as homocysteinemia over 15 mol/l, cigarette smoking), family history of pre-eclampsia/eclampsia and/or of cardiovascular predisposing factors (as above), presence of rheumatological and/or immunological disorders, pre-existing thrombophilia.
  Maternal only: history of pre-eclampsia, over 10 years from last pregnancy, multiple partners, assisted reproductive technology (ART), oocyte or embryo donation, weight at term (Kg).

SECONDARY OUTCOMES:
Maternal outcomes measured by a novel multiple choice on-line questionnaire | Three months
  gestational week at term; gestational diabetes (defined as fasting plasma glucose level over 126 mg/dl or a fasting glycemia over 92 mg/dl and a 1-hour glycemia over 180 mg/dl and a 2-hour glycemia over 153 mg/dL in the 75 g oral glucose tolerance test), hypertension (defined as a diastolic blood pressure ≥ 90 mm Hg and a systolic blood pressure ≥ 140 mmHg on at least two different recordings taken at least 4-6 h apart and less than 7 days apart, using an appropriate cuff) and/or kidney failure (defined by the abrupt loss of kidney function; a serum creatinine concentration above 0.8 mg/dL during pregnancy may indicate an underlying renal dysfunction) resolved after childbirth or within 3 months from delivery or over 3 months from delivery or current.
Fetal outcomes measured by a novel multiple choice on-line questionnaire | Three months
  weight at birth (grams), blood group when tested, abortion

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Viviani, M.D., Principal Investigator — ASST Papa Giovanni XXIII, Bergamo, Italy
Locations (1):
- Asst Papa Giovanni Xxiii, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: Undecided